CLINICAL TRIAL: NCT06683833
Title: Comparative Analysis of Egyptian MTA, Biodentine, and Calcium Hydroxide as Indirect Pulp Capping Materials in Permanent Teeth. (A 6m Randomized Clinical Trial)
Brief Title: Comparison Between Egyptian MTA, Biodentine Versus Calcium Hydroxide as Indirect Pulp Capping Materials In Permanent Teeth
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Talaat Mostafa Elsorogy, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: operative 2
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Deep Caries; Indirect Pulp Capping; Mineral Trioxide Aggregate (MTA); Calcium Hydroxide; Biodentine; Patient Reported Outcome Measures
Keywords: Deep caries; Indirect pulp capping; Mineral trioxide aggregate (MTA); Calcium hydroxide; Biodentine; Patient reported outcomes measures (PROMS); Randomized clinical trial
MeSH Terms: interventions — tricalcium silicate; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: * Outcome assessors and analyst will be blinded to the intervention group assigned to the patients.
  * Participants will be blinded from knowing the material used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Egyptian MTA (Experimental): * Complete caries removal from the cavity.
  * The liquid of Egyptian MTA (Toothmate) will be mixed with powder according to the manufacturers' instructions.
  * The capping materials will be placed with the passive application on the deepest part of the cavity. Only light pressure will be applied on the MTA mixture using a wet cotton pellet to ensure adaptation of the material onto the dentin.
  * A light-cured glass ionomer cement base will be applied in the cavity .
  * Selective enamel etching will be applied on enamel only.
  * The one-bottle universal adhesive system bond will be applied on enamel and dentine.
  * A Nano hybrid composite resin material will then be incrementally inserted into the cavities.
  Interventions: Drug: Egyptian MTA
- Biodentine (Experimental): * Complete caries removal from the cavity.
  * Gently tapping a capsule of Biodentine (Septodont) on a hard surface to loosen the powder, then opening the capsule, Detaching a single-dose container of liquid and gently tapping on the sealed cap to force all the liquid down the container, Twisting cap to open, Then Pouring 5 drops from the single-dose container into the capsule, Then Closing the capsule and Placing it on a mixing device for 30 seconds, Then Collecting Biodentine with the instrument supplied in the box.
  * The capping materials will be placed with the passive application on the deepest part of the cavity.
  * A light-cured glass ionomer cement base will be applied in the cavity .
  * Selective enamel etching will be applied on enamel only.
  * The one-bottle universal adhesive system bond will be applied on enamel and dentine.
  * A Nano hybrid composite resin material will then be incrementally inserted into the cavities.
  Interventions: Drug: Biodentine
- Calcium Hydroxide (Active Comparator): * Complete caries removal from the cavity.
  * According to the manufacturers' instructions, Dispensing equal volumes of base and catalyst pastes on the parchment paper pad provided. Using a Dycal (Dentsply) Liner applicator, stirring immediately to mix thoroughly until a uniform color is achieved, complete mixing occurs within 10 seconds, using the ball-pointed Dycal Liner applicator or similar instrument, the mix will be placed directly on the cavity.
  * The capping materials will be placed with the passive application on the deepest part of the cavity.
  * A light-cured glass ionomer cement base will be applied in the cavity .
  * Selective enamel etching will be applied on enamel only.
  * The one-bottle universal adhesive system bond will be applied on enamel and dentine.
  * A Nano hybrid composite resin material will then be incrementally inserted into the cavities.
  Interventions: Drug: Calcium Hydroxide (Ca(OH)2)

INTERVENTIONS:
Drug: Egyptian MTA — * Complete caries removal from the cavity.
  * The liquid of Egyptian MTA (Toothmate) will be mixed with powder according to the manufacturers' instructions.
  * The capping materials will be placed with the passive application on the deepest part of the cavity. Only light pressure will be applied on the MTA mixture using a wet cotton pellet to ensure adaptation of the material onto the dentin.
  * A light-cured glass ionomer cement base will be applied in the cavity .
  * Selective enamel etching will be applied on enamel only.
  * The one-bottle universal adhesive system bond will be applied on enamel and dentine.
  * A Nano hybrid composite resin material will then be incrementally inserted into the cavities.
  Arms: Egyptian MTA
Drug: Biodentine — * Complete caries removal from the cavity.
  * Gently tapping a capsule of Biodentine (Septodont) on a hard surface to loosen the powder, then opening the capsule, Detaching a single-dose container of liquid and gently tapping on the sealed cap to force all the liquid down the container, Twisting cap to open, Then Pouring 5 drops from the single-dose container into the capsule, Then Closing the capsule and Placing it on a mixing device for 30 seconds, Then Collecting Biodentine with the instrument supplied in the box.
  * The capping materials will be placed with the passive application on the deepest part of the cavity.
  * A light-cured glass ionomer cement base will be applied in the cavity .
  * Selective enamel etching will be applied on enamel only.
  * The one-bottle universal adhesive system bond will be applied on enamel and dentine.
  * A Nano hybrid composite resin material will then be incrementally inserted into the cavities.
  Arms: Biodentine
Drug: Calcium Hydroxide (Ca(OH)2) — * Complete caries removal from the cavity.
  * According to the manufacturers' instructions, Dispensing equal volumes of base and catalyst pastes on the parchment paper pad provided. Using a Dycal (Dentsply) Liner applicator, stirring immediately to mix thoroughly until a uniform color is achieved, complete mixing occurs within 10 seconds, using the ball-pointed Dycal Liner applicator or similar instrument, the mix will be placed directly on the cavity.
  * The capping materials will be placed with the passive application on the deepest part of the cavity.
  * A light-cured glass ionomer cement base will be applied in the cavity .
  * Selective enamel etching will be applied on enamel only.
  * The one-bottle universal adhesive system bond will be applied on enamel and dentine.
  * A Nano hybrid composite resin material will then be incrementally inserted into the cavities.
  Arms: Calcium Hydroxide

SUMMARY:
Compare the clinical performance and patient satisfaction of Egyptian MTA, Biodentine versus Calcium Hydroxide as indirect pulp capping materials in permanent teeth

DETAILED DESCRIPTION:
Vital pulp treatments (VPTs) represent a group of minimally invasive treatments intended to preserve the health of all or part of the dental pulp. These treatments include a spectrum of modalities including indirect pulp capping as first option, direct pulp capping and pulpotomy (partial or complete).

Indirect pulp capping (IPC) has been proposed as a conservative pulp therapy for several decades. It is a technique for deep caries management without any features of pulp degeneration.This stimulates tertiary dentin formation, avoiding pulp exposure and maintaining pulp vitality. Cases of indirect pulp capping in deep cavities are those where the residual dentin thickness is equal or less than 0.5 mm, the number and size of the "open" dentinal tubules are such that communication with the pulp parenchyma is comparable to that of a true exposure.

Ideal pulp capping material should maintain pulpal vitality and stimulate reparative dentin formation. These materials should possess certain properties such as biocompatibility, bioactivity, radiopacity, insolubility, dimensional stability, and adequate adhesive ability to both the dentin and to the restorative materials. It should also release remineralizing ions, provide bacterial seal, prevent secondary caries, should have bactericidal or bacteriostatic activity against the causative pathogens, and promote the formation of mineralized tissue

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 22: 45 years old.
* Males or females.
* Patients with vital teeth with deep carious lesions.
* Patients in good general health.
* Good oral hygiene.
* Co-operative patients who show interest to participate in the study.

Exclusion Criteria:

* Patients with systemic diseases.
* Patients with known allergic or adverse reaction to the tested materials.
* Patients with bad oral hygiene.
* Patient who frequently use analgesic or any drugs that could mask the pain.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of treatment success | T( Time) T0( base line)= one week after , T2= 3 months , T3= 6 months
  Pulp response to different stimuli by thermal and electrical pulp tests. When tooth normally responds to thermal and electrical pulp tests = success When tooth doesn't respond to thermal and electrical pulp tests = failure

SECONDARY OUTCOMES:
Clinical assessment of pain | T( time) T0( baseline )= 1 week after, T1= 3 months, T2= 6 months
  Patient reported outcome measures by visual analogue scale visual analogue scale is used to describe the pain by patients themselves in scores as ( 0: no pain ) & (7-10 : Severe pain)
Patient satisfaction with the treatment | T( time) T0= 1 week after, T1= 3 months , T2= 6 months
  Patient reported outcome measure by 4- point likert scale 4- point likert scale used to describe patient satisfaction with the treatment as " (a) yes, very satisfied" & " (d) not all satisfied"